CLINICAL TRIAL: NCT03434314
Title: Paraplegia Prevention in Aortic Aneurysm Repair by Thoracoabdominal Staging With 'Minimally-Invasive Segmental Artery Coil-Embolization': A Randomized Controlled Multicentre Trial - PAPAartis
Brief Title: Paraplegia Prevention in Aortic Aneurysm Repair by Thoracoabdominal Staging
Acronym: PAPAartis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: European Commission (Other); German Research Foundation (Other); Universidad de Granada (Other); European Clinical Research Infrastructure Network (Other); Modus Research and Innovation Limited (Unknown); Rigshospitalet, Denmark (Other); European Society of Cardiology (Network); Baylor College of Medicine (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, David Petroff, Dr. David Petroff [Prof. Dr. Christian Etz], University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAPAartis; 733203 (Other Grant/Funding Number: Horizon2020, European Commission); ET 127/2-1 (Other Grant/Funding Number: German Research Foundation)
Record Dates: First submitted 2018-01-12; First posted 2018-02-15 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Aortic Aneurysm, Thoracoabdominal
Keywords: Paraplegia; Aortic Aneurysm Repair; Staging; Embolization; TAAA; Thoracoabdominal aortic aneurysm; MISACE; Spinal cord ischemia; Spinal cord ischaemia; Spinal cord injury; Spinal cord ischemic injury; Spinal cord ischaemic injury; Permanent paraplegia; Temporary paraplegia; Paraparesis; SCI; TAAA repair; Open TAAA repair; Open surgical TAAA repair; Endovascular TAAA repair; TEVAR; Aortic surgery; Thoracoabdominal aortic surgery; Type B aortic dissection; Chronic type B aortic dissection; Stanford type B aortic dissection; Collateral network; Paraspinal collateral network; Paraspinous collateral network; Arteriogenesis; Intercostal arteries
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Paraplegia; Spinal Cord Ischemia; Spinal Cord Injuries; Paraparesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MISACE arm (Experimental): Minimally-Invasive Segmental Artery Coil-Embolization
  MISACE procedure prior to aneurysm repair
  segmental arteries are occluded with coils or plugs in one to three MISACE sessions (staged procedure)
  Interventions: Procedure: Minimally-Invasive Segmental Artery Coil-Embolization
- control arm (No Intervention): receives treatment of aneurysm as usual: open surgical repair or endovascular repair without MISACE

INTERVENTIONS:
Procedure: Minimally-Invasive Segmental Artery Coil-Embolization — During one single MISACE session 3-7 segmental arteries will be occluded. The procedure is conducted through a peripheral artery access in local anaesthesia. Microcoils or vascular plugs will be used for the occlusion itself.
  Arms: MISACE arm

SUMMARY:
Aortic aneurysms represent the most common and dangerous aortic diseases. Although conventional aortic repair techniques cure the disease, there is a high risk of paraplegia particularly in extensive thoracoabdominal aneurysms due to impaired blood supply to the spinal cord.

The PAPA-ARTiS trial will assess the clinical safety and efficacy of the MISACE (Minimally-Invasive Segmental Artery Coil-Embolization) procedure, a novel therapeutic concept to reduce the risk of paraplegia due to aneurysm repair.

The study investigates the MISACE procedure as a potential pre-treatment prior to open or endovascular aneurysm repair in patients with thoracoabdominal aortic aneurysms. Patients will be randomized to one of the two treatment strategies: a) aneurysm repair without MISACE pre-treatment, or b) aneurysm repair with MISACE pre-treatment.

DETAILED DESCRIPTION:
Chronic aortic aneurysms are permanent and localized dilations of the aorta that remain asymptomatic for long periods of time, but continue to increase in diameter before they eventually rupture. Left untreated, the patients' prognosis is dismal, since the internal bleeding of the rupture brings about sudden death. Although successful treatment cures the disease, the risky procedures compromise spinal cord blood supply acutely and permanently, frequently leading to paraplegia, particularly for aneurysms involving crucial segmental arteries, i.e. thoracoabdominal aortic aneurysms of Crawford type II & III. Although various strategies have achieved a remarkable decrease in the incidence of paraplegia, it is still no less than 10-20%.

However, it has recently been found that the deliberate staged occlusion of the segmental arteries to the paraspinous collateral network finally supplying the spinal cord can trigger arterial collateralization, thus stabilizing blood supply from alternate inflow sources and preventing ischaemia.

This has been translated to a clinically available therapeutic option, 'minimally invasive staged segmental artery coil embolization' (MISACE), which proceeds in a 'staged' manner to occlude groups of arteries under highly controlled conditions, after which time must be allowed for arteriogenesis to build a robust collateral blood supply.

PAPA-ARTiS is a multi-national, prospective, open-label, two-arm, randomized controlled trial to demonstrate, that a minimally invasive staged treatment approach can reduce paraplegia and mortality in patients undergoing thoracoabdominal aortic aneurysm (TAAA) repair.

Patients with planned aneurysm repair will be included in the study and will be randomized 1:1 in the control group or the MISACE-group. The control group receives treatment as per standard institutional protocol - open or endovascular repair without MISACE. In the MISACE-group, segmental arteries will be occluded in one to three sessions some weeks before the definite repair. Segmental arteries are occluded with coils or plugs.This induces arteriogenesis and the building of a robust collateral network ultimately supplying the spinal cord. During aneurysm repair, these new arteries provide an alternate blood supply to the spinal cord and thereby help prevent paraplegia.

ELIGIBILITY:
Inclusion Criteria:

* TAAA, Crawford type II or III
* planned open or endovascular repair of aneurysm within four months
* ≥ 18 years old

Exclusion Criteria:

* complicated (sub-) acute type B aortic dissection
* ruptured and urgent aneurysm (emergencies)
* untreated aortic arch aneurysm
* bilaterally occluded iliac arteries or chronic total occlusion of left subclavian artery
* pre-operative neurological deficits or spinal cord dysfunction
* major untreated cardio-pulmonary disease
* life-expectancy of less than one year
* high risk for segmental artery embolism
* severe contrast agent allergy, severe reduction in glomerular filtration rate (CKD stage 4)
* expected lack of compliance
* pregnant or nursing women
* impaired thyroid function, if not under stable treatment
* women of child bearing potential without highly effective contraceptive measures
* current participation in other interventional clinical trial
* patients under legal supervision or guardianship
* patients placed in an institution by official or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-11-08 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to greatly reduce incidence of ischaemic spinal cord injury and mortality. | 30 days after TAAA repair
  Successful treatment of the aneurysm is a binary variable. All of the following criteria must be met for this composite endpoint to count as a success:
  * The patient is alive and without substantial spinal cord injury 30 days after treatment, and
  * the aneurysm did not rupture and has been excluded within six months of randomization. Substantial spinal cord injury will be determined with a modified Tarlov scale (see below).

SECONDARY OUTCOMES:
substantial spinal cord injury | 30 days after TAAA repair and at one year after TAAA repair
  Substantial spinal cord injury is defined as zero to two on the modified Tarlov scale.
  0. No lower extremity movement
  1. Lower extremity motion without gravity
  2. Lower extremity motion against gravity
  3. Able to stand with assistance
  4. Able to walk with assistance
  5. Normal
spinal cord injury according to the modified Tarlov scale from TAAA repair to one year | from date of TAAA repair and up to one year after TAAA repair
  Spinal cord injury will be determined with a modified Tarlov scale (see above).
mortality | at 30 days and one year after TAAA repair
  all-cause mortality
stay in intensive care unit and intermediate care | from date of TAAA repair and up to one year after TAAA repair
  length of stay in intensive care unit and intermediate care unit after TAAA repair
sub-group analyses | up to one year after TAAA repair
  sub-group analyses of spinal cord injury according to modified Tarlov scale (see above) for open repair and endovascular repair separately
sub-group analyses | up to one year after TAAA repair
  sub-group analyses of mortality for open repair and endovascular repair separately
re-operation for bleeding | from date of TAAA repair and up to one year after TAAA repair
  re-operation for bleeding (only for open repair)
cross-clamping times | during open surgery
  cross-clamping times during open surgery
residual aneurysm sac perfusion | up to one year after TAAA repair
  residual aneurysm sac perfusion, i.e. type II endoleaks (only for endovascular repair)
costs | up to one year after TAAA repair
  incremental cost-effectiveness ratio (ICER) will be calculated
Quality Adjusted Life Years | up to one year after TAAA repair
  Quality Adjusted Life Years (QALYs) will be estimated over one year

CONTACTS AND LOCATIONS:
Overall Officials: Christian D Etz, Prof. Dr., Principal Investigator — University Leipzig
Locations (29):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Herzzentrum Hietzing, Vienna
- France (2):
  - University Hospital of Bordeaux, Bordeaux
  - Marie Lannelongue Hospital, Le Plessis-Robinson
- Germany (16):
  - Uniklinik RWTH Aachen, Aachen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Westdeutsches Herz und Gefäßzentrum Essen, Essen
  - Universitäts-Herzzentrum Freiburg/ Bad Krozingen, Freiburg im Breisgau
  - Herzzentrum Hamburg, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Herzzentrum Leipzig, Leipzig
  - UniversitätskIinikum Leipzig, Leipzig
  - Klinikum rechts der Isar (TU München), Munich
  - Klinikum der Universität München (LMU), München
  - Universitätsklinikum Münster, Münster
  - Paracelsus Universität - Klinikum Nürnberg, Nuremberg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Italy (2):
  - S.Orsola-Malpighi Hospital, Bologna
  - Ospedale San Raffaele SRL, Milan
- Maastricht University Medical Center, Maastricht, Netherlands
- Poland (2):
  - Medical University of Warsaw, Warsaw
  - Silesian Center for Heart Diseases, Zabrze
- Sweden (2):
  - Lund University Hospital Malmoe, Malmo
  - Örebro University Hospital, Örebro
- Bern University Hospital, Bern, Switzerland
- St Bartholomews Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Petroff D, Czerny M, Kolbel T, Melissano G, Lonn L, Haunschild J, von Aspern K, Neuhaus P, Pelz J, Epstein DM, Romo-Aviles N, Piotrowski K, Etz CD. Paraplegia prevention in aortic aneurysm repair by thoracoabdominal staging with 'minimally invasive staged segmental artery coil embolisation' (MIS(2)ACE): trial protocol for a randomised controlled multicentre trial. BMJ Open. 2019 Mar 4;9(3):e025488. doi: 10.1136/bmjopen-2018-025488. PMID 30837256